CLINICAL TRIAL: NCT04968119
Title: A Novel Telehealth Exercise Platform to Reduce Frailty in Hematopoietic Cell Transplantation Survivors: A Pilot Feasibility Study
Brief Title: Telehealth Exercise Platform to Reduce Frailty After Bone Marrow Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20731; NCI-2021-03539 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20731 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-07-20 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (telehealth intervention) (Experimental): Patients participate in telehealth exercise sessions at home over 30 minutes with a trainer 3 days a week for 8 weeks (24 total sessions).
  Interventions: Other: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (delayed exercise intervention) (Active Comparator): Patients maintain their normal activities of daily living for 8 weeks before participating in the telehealth exercise program as described in Arm I.
  Interventions: Other: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Exercise Intervention — Participate in telehealth exercise sessions
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the feasibility of implementing a telehealth exercise platform to reduce frailty in patients after bone marrow transplant.

The exercise program uses a telehealth platform (e.g. smart phones, tablets or computers) to view pre-recorded exercise videos on coordination, posture, stretching, balance and resistance/aerobic training.

Physical activity may help to improve physical function, including frailty, after bone marrow transplant. Information from this trial may help researchers design future telehealth exercise routines for treating people with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of the telehealth exercise program, as evaluated by participation and completion rates.

SECONDARY OBJECTIVE:

I. Explore the effects of the telehealth exercise program on physical functioning.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients participate in telehealth exercise sessions at home over 30 minutes with a trainer 3 days a week for 8 weeks (24 total sessions).

ARM B: Patients maintain their normal activities of daily living for 8 weeks before participating in the telehealth exercise program as described in Arm I.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age at the time of study enrollment
* >= 2-years from hematopoietic cell transplantation (HCT) and in clinical remission
* Identified as pre-frail or frail based on Bone Marrow Transplant Survivorship Study (BMTSS) questionnaire (i.e. clinically underweight, exhaustion, low energy expenditure, slow walking speed, and muscle weakness), with the presence of >= 3/5 indices classified as frail and 2/5 indices classified as prefrail
* Able to understand and sign the informed consent document
* Physically able and willing to complete all study procedures
* Has access to the internet and a smartphone
* English speaking

Exclusion Criteria:

* Overt cardiovascular disease (e.g. myocardial infarction, stroke, angina)
* Contraindications to exercise (acute infectious disease, physical disability preventing safe performance [assistive devices], cognitive impairment or inability to cooperate)
* Participation in regular exercise (> 60 minutes per week)
* Female who are pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Participation rate | Week 9
  Rate of participation is defined as number of hematopoietic cell transplantation (HCT) survivors who were approached and participated divided by the total number of eligible HCT survivors who were approached for the study and then multiplied by 100%.
  Will be considered feasible if >= 50% of eligible patients that are approached for participation enroll onto the study.
  Minimal descriptive statistical analyses will be performed for all participant baseline characteristics and compared across groups to test for balance across the groups, using t-tests (or non-parametric Wilcoxon rank sum) for continuous variables and chi-square tests for categorical variables.
Intervention completion rate | Week 9
  Will be considered feasible if >= 75% of enrolled participants successfully complete all study measurements (remote physical function) and > 50% of patients randomized to the intervention arm are able to complete > 70% of total exercise sessions (17/24 sessions).
  Minimal descriptive statistical analyses will be performed for all participant baseline characteristics and compared across groups to test for balance across the groups, using t-tests (or non-parametric Wilcoxon rank sum) for continuous variables and chi square tests for categorical variables.

SECONDARY OUTCOMES:
Changes in the efficacy of the telehealth exercise program on physical functioning - Timed balance | From baseline to week 9
  Physical functioning (Timed balance) will be measured in the unit of time as seconds.
Changes in the efficacy of the telehealth exercise program on physical functioning - Gait speed | From baseline to week 9
  Physical functioning (Gait speed ) will be measured in the unit of time as seconds.
Changes in the efficacy of the telehealth exercise program on physical functioning - Chair stand | From baseline to week 9
  Physical functioning (Chair stand ) will be measured in the unit of time as seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Kyuwan Lee, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Lee K, Shamunee J, Lindenfeld L, Ross E, Hageman L, Sedrak MS, Wong FL, Nakamura R, Forman SJ, Bhatia S, Armenian SH. Feasibility of implementing a supervised telehealth exercise intervention in frail survivors of hematopoietic cell transplantation: a pilot randomized trial. BMC Cancer. 2023 May 1;23(1):390. doi: 10.1186/s12885-023-10884-5. PMID 37127595